CLINICAL TRIAL: NCT01125878
Title: Understanding Resistant Starch on Satiety in Premenopausal Women
Brief Title: Types of Resistant Starch and Their Effect on Appetite
Acronym: NST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NST 2010-027
Record Dates: First submitted 2010-05-11; First posted 2010-05-19 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Psychological Phenomena and Processes
Keywords: satiety; appetite; fiber; starch; nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Starch Composite B (Active Comparator): fiber mixture
  Interventions: Dietary Supplement: Starch composite B
- Starch Composite C (Active Comparator): fiber mixture
  Interventions: Dietary Supplement: Starch composite C
- Starch Composite D (Active Comparator): fiber mixture
  Interventions: Dietary Supplement: Starch composite D
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — placebo
  Arms: Placebo
Dietary Supplement: Starch composite B — fiber mixture
  Arms: Starch Composite B
Dietary Supplement: Starch composite C — fiber mixture
  Arms: Starch Composite C
Dietary Supplement: Starch composite D — fiber mixture
  Arms: Starch Composite D

SUMMARY:
Investigators are interested in learning how appetite responds to certain types of starch and fiber mixtures. In this research study, subjects will be asked to consume cookie bars containing different types of starch and fiber mixtures, then describe their feelings of hunger, fullness and desire to eat for the 3 hour study period. Subjects will be asked to do this on four separate occasions. Following the 3 hour study period, a deli-style lunch will be served. Investigators want to see how appetite responds to these four different starch and fiber mixtures.

DETAILED DESCRIPTION:
This study will require one initial screening visit (approximately 1 hour) and four study visits each lasting approximately 4 hours. All visits should be done in 2 months. We are looking for healthy, non-smoking, premenopausal female volunteers older than 18 with no medical history of diabetics, heart, lung, kidney, stomach, or liver disease.

The initial screening visit will determine subject eligibility through height, weight and waist circumference measurements, blood glucose finger prick and eating, health and mood surveys.

If willing and eligible to participate, subjects will have four study visits. All study visits will be scheduled according to each individual subject's menstrual cycle. At each visit subject will be asked to eat the cookie bar and then answer questions about their feelings of hunger, fullness and desire to eat. Subject will continue to answer questions about their feelings of hunger, fullness and desire to eat at specific time points up to 3 hours after eating the yogurt. After 3 hours a lunch meal will be served. The lunch meal consists of typical deli items, such as pasta, rolls, salad, etc. Subject will be allowed to eat as much or as little of the lunch as they'd like.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females
* 18 years of age and older
* BMI (body mass index) between 18.5 and 24.9 kg/m2 inclusive
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* unrestrained eater (score < 10 on the Three Factor Eating Questionnaire)

Exclusion Criteria:

* Pregnant and/or lactating or planning for pregnancy
* Allergies or intolerances to foods consumed in the study
* Fasting blood glucose > 110 mg/dL. Subjects identified with elevated fasting blood glucose levels will be will be advised to contact their primary care physician for appropriate follow-up care.
* Taking over the counter fiber supplements or other supplements that may interfere with the study procedures or endpoints
* Taking prescription medications that may interfere with study procedures or endpoints (medications that affect appetite)
* Subjects with unusual dietary habits (e.g. pica)
* Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 kg in a 60 day period)
* Excessive exercisers or trained athletes
* Addicted to drugs and/or alcohol
* Medically documented psychiatric or neurological disturbances
* Smoker (past smoker may be allowed if cessation is > 2 years)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09-02 (Actual); Primary Completion 2011-07-12 (Actual); Study Completion 2011-09-29 (Actual)

PRIMARY OUTCOMES:
Subjective and behavioral satiety responses after consumption of the resistant starch composites by visual analog scales and subsequent food intake. | 3 hour postprandial study
  Meals will be provided under fasting conditions and thereafter subjects will record satiety reponses at 30 mins, 60, 90, 120, 150 and 180 on a visual analog scale (VAS). The subject will answer a series of questions on the VAS describing their feelings of hunger, fullness and desire to eat at the above mentioned time points.
  Satiety will also be determined on the quantity of the test lunch meal consumed. This test meal will be served three hours after consumption of the starch composites.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, PhD, MS, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology; Indika Edirisinghe, PhD, Principal Investigator — Clinical Nutrition Research Center, Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robertson MD, Currie JM, Morgan LM, Jewell DP, Frayn KN. Prior short-term consumption of resistant starch enhances postprandial insulin sensitivity in healthy subjects. Diabetologia. 2003 May;46(5):659-65. doi: 10.1007/s00125-003-1081-0. Epub 2003 Apr 24. PMID 12712245
- [Background] Robertson MD, Bickerton AS, Dennis AL, Vidal H, Frayn KN. Insulin-sensitizing effects of dietary resistant starch and effects on skeletal muscle and adipose tissue metabolism. Am J Clin Nutr. 2005 Sep;82(3):559-67. doi: 10.1093/ajcn.82.3.559. PMID 16155268